CLINICAL TRIAL: NCT03562325
Title: Acceptance & Commitment Therapy for ME/CFS (Chronic Fatigue Syndrome) - an Open Case Trial
Brief Title: ACT for ME/CFS - an Open Case Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rikard Wicksell (Other)
Collaborators: Region Stockholm (Other Government); Skandia Insurance Company, Ltd. (Unknown)
Responsible Party: Sponsor-Investigator, Rikard Wicksell, Associate Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015/370-31/4
Record Dates: First submitted 2018-06-08; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Chronic Fatigue Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Open case trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACT (Other): Acceptance & Commitment Therapy (ACT)
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — The main target in ACT for ME/CFS (as for Fibromyalgia and Chronic pain in previous studies by our group) is to promote a shift of perspective in life from symptom reduction (when it does not work) to a valued life. As such it entails acceptance and exposure to discomfort, in order to lessen the effects of negative experiences (symptoms, emotions, thoughts) on behaviours in everyday life.

SUMMARY:
The goal of this research project is to evaluate if our well-researched behavior medicine treatment model for chronic pain, based on Acceptance and Commitment Therapy, is safe and effective in increasing quality of life and functioning also in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS). To date there are no effective treatments for ME/CFS as the ethology and pathophysiology are unknown, while levels of functioning and quality of life as well as secondary effects such as depressive and anxiety symptoms indicate a highly affected patient population. As such, there is a need for behavior medicine approaches that aim to alleviate suffering and promote increases in quality of life for these patients. The aim of the present study is to do a preliminary evaluation of the safety, acceptability and efficacy of an ACT-based treatment protocol for ME/CFS. An additional aim is to explore potential mediators of change for the effect of treatment on disability.

DETAILED DESCRIPTION:
Background Medical strategies alone appear insufficient to increase functioning and quality of life in ME/CFS. Cognitive behavioral therapy (CBT) is the only treatment approach with preliminary evidence of efficacy for improving functioning and quality of life. However, effect sizes are generally modest.

Behavior medicine treatment approaches based on Acceptance & Commitment Therapy (ACT) have gained increasing attention and research support within clinical trials for similar diagnoses (e.g. chronic pain, Fibromyalgia). Results from these areas illustrate the utility of this approach for individuals with somatic symptomatology. To date, the efficacy of ACT has not been evaluated for ME/CFS.

Purpose The aims of this pilot study are to explore the utility of ACT and to evaluate the feasibility of the treatment model for patients with ME/CFS.

Method Treatment program: 13 weekly to bi-weekly individual ACT sessions with a psychologist (10) and a physician (3) respectively.

An open trial design is used, with assessments at pre-, mid- and post-treatment as well as at 3 and 6 months follow-up. Further, yearly follow-ups until 5-year follow-up are planned.

Measures: History data, illness factors, psychological factors, functioning and quality of life.

Patients: Consecutively recruited via referrals to a specialist treatment centre (n=40). Once patients have been found eligible and expressed interest in study participation they will be assessed by a psychologist and by a physician, via semi-structured interviews to confirm eligibility and to ensure that the patient meet the study criteria. Informed consent is obtained from all participants prior to the assessment.

Statistical analysis: Evaluations of treatment effects are primarily based on intent-to-treat analyses. The statistical approach will primarily be based on linear multilevel modeling (LMM), which takes into account dependencies between repeated measures and differences between patients in pre-treatment status and treatment response (i.e. random effects modeling) and also provide means of handling missing data.

ELIGIBILITY:
Inclusion Criteria: Subjects were included if

* Referred to a specialist behavior medicine treatment unit for ME/CFS
* 18 years of age or older
* Fulfilling CDC ME/CFS diagnostic criteria AND 2003 clinical case definition ME/CFS diagnostic criteria
* Treatment resistent symptomatology
* Evident ME/CFS-related disability (assessed with self-report questionnaires and clinical interviews)
* Stabile medication during the last 2 months with no planned changes during active study treatment

Exclusion Criteria: Subjects were excluded if:

* psychiatric or somatic comorbidity was prevalent and assessed as more primary than ME/CFS illness;
* non-adherence during assessment phase;
* they did not speak Swedish;
* ongoing or recently (less than six months) completed CBT-oriented treatment;
* other treatment than standard care (pharmacological, psychological or otherwise) planned in the coming six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-11-10 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
ME/CFS Disability Index (changes between assessments) | Baseline to 6-month follow-up
  Self-reported ME/CFS-related disability in 7 life domains (domestic; recreational activities; social activities; occupational; sexual life; daily activities; life-sustaining activities). Each item is scored 0-10 (0= no disability, 10=total disability).
Psychological Inflexibility in Fatigue Scale (PIFS) (changes between assessments) | Baseline to 6-month follow-up
  Self-rated psychological inflexibility related to fatigue

SECONDARY OUTCOMES:
ME/CFS Symptoms (changes between assessments) | Baseline to 6-month follow-up
  Self-reported prevalence and intensity (0-4) of ME/CFS symptoms based on the 2003 clinical case definition (0=symptom absence, 4=unbearable).

CONTACTS AND LOCATIONS:
Overall Officials: Rikard Wicksell, PhD, Study Director — Director of Functional Area Medical Psychology, Karolinska Univ Hospital, assoc professor and head of research group Behavior Medcine, Karolinska Institutet, Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No